CLINICAL TRIAL: NCT06866587
Title: Evaluation of Proprioceptive Sense in Patients With Acute Non-specific Neck Pain and Elucidation of Its Relationship With Cervical Vertigo.
Brief Title: Cervical Dizziness in Patients With Acute Non-specific Neck Pain
Acronym: dizziness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Semra Ağırbaş, asst.prof.dr, Yuzuncu Yil University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04.04.2019/ 2019-07
Record Dates: First submitted 2025-02-27; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Dizziness; Neck Pain; Elastography
Keywords: elastography; neck pain; cervical dizziness
MeSH Terms: conditions — Dizziness; Neck Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: A number of questionnaires were administered to the patients, including Demographic Data Form, Neck Pain Visual Analogue Scale (Neck-VAS), Neck Disability Index (NDI), Dizziness Handicap Inventory (DHI), Dizziness Visual Analogue Scale (Dizziness-VAS), Vertigo Dizziness Imbalance Symptom Scale (VDI-SS), and Quality of Life Scale (VDI-QOLS) both before and after treatment. Patients that had a recurrent attack of CD during the follow-up period underwent shear-wave elastography (SWE) for the assessment of the stiffness of neck muscles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients diagnosed with cervical dizziness (Other): A patient-specific, comprehensive clinical examination was performed in each patient. In addition, a detailed patient history was obtained from each patient. To diagnose CD, Head- Neck Differentiation Test (HNDT) and Cervical Torsion Test (CTT) were performed using Frenzel lenses. Patients that were found to be positive in either of these two tests after the exclusion of other peripheral and central causes were diagnosed with cervical Dizziness.
  Interventions: Other: exercise therapy

INTERVENTIONS:
Other: exercise therapy — Priorities of the treatment included care and interventions to avoid inappropriate neck positions and to provide a regular exercise program for neck muscles and ergonomics training (ergonomic arrangements for desk setup, reading position, computer and mobile phone use, handcrafts, television watching, and pillow height). Of note, patients were advised to avoid cold exposure, particularly in the neck area (air-conditioned environments, wet hair, and holding the hair dryer too close to the scalp). Patients that did not show improvement after training and regular exercise were initiated on medical treatment after the second week and were given myorelaxant gel and oral tablets (diclofenac sodium) for the neck area.

SUMMARY:
Acute non-specific neck pain (ANSNP) is one of the causes of cervicogenic dizziness (CD).To investigate the severity of CD in patients with ANSNP and to determine the efficacy of the treatment and follow-up.

DETAILED DESCRIPTION:
The primary aim of this study was to investigate the contribution of cervical proprioception impairment to the development of cervical dızzıness in patients with acute non specific neck pain and to determine the efficacy of the treatment and follow-up performed in patients coexisting with cervical dizziness and nonspecific neck pain. Our hypothesis was that the objective measurement of muscle stiffness with shear-wave elastography could aid in the differential diagnosis in patients coexisting with cervical dizziness and non specific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were as follows: pain on palpation in the neck area, neck stiffness, tension and tenderness in the neck muscles, and cervical movement limitation. All the patients included in the study had no history of a maneuver for dizziness, no history of ototoxic drug use, and had normal hearing.

Exclusion Criteria:

* Exclusion criteria included presence of benign paroxysmal positional vertigo (BPPV), Meniere's disease, migraine-associated vertigo, vertebrobasilar insufficiency, postural hypotension, a history of trauma to the cervical region, myofascial pain syndrome, and neurological, rheumatological, and systemic diseases. Additionally, patients detected with neck-related conditions (cervical spondylosis, cervical disc hernia, fracture, dislocation, spondylolisthesis, scoliosis) and fibromyalgia in cervical magnetic resonance imaging (MRI) were also excluded from the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2019-04-14 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Neck pain Visual analog scale scores | Patients were invited for follow-up visits at 2, 6, 8 weeks and at 3, 4, 6, and 12 months.
  Neck Pain Visual Analogue Scale (Neck-VAS) consists of an 11-point numerical rating scale, in which 0 indicates "no pain at all" and 10 indicates "worst possible pain."
Dizziness Handicap Inventory, | Patients were invited for follow-up visits at 2, 6, 8 weeks and at 3, 4, 6, and 12 months.
  Disability Index (NDI), developed as a modification of the Oswestry Disability Index, was used to assess neck pain-specific disability. NDI consists of 10 items including (i) pain, (ii) personal care, (iii) lifting, (iv) reading, (v) headaches, (vi) concentration, (vii) work, (viii) driving, (ix) sleeping, and (x) recreation. Each item is rated on a 6-point Likert scale (0= no disability, 5= total disability) and the scoring intervals for interpretation include 0-4 (no limitation), 5-14 (mild limitation), 15-24 (moderate limitation), 25-34 (severe limitation), and above 34 (completely limited).
Vertigo Dizziness Imbalance Symptom Scale (VDI-SS), | Patients were invited for follow-up visits at 2, 6, 8 weeks and at 3, 4, 6, and 12 months.
  Vertigo Dizziness Imbalance Symptom Scale (VDI-SS) is used to assess head imbalance and the severity and frequency of dizziness symptoms. The scale consists of 14 items scored between 0 and 5. Vertigo Dizziness Imbalance Quality of Life Scale (VDI- QOLS) consists of 22 items scored between 0 and 5 and the severity of the symptoms is evaluated based on the total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Yüzüncü yıl University Faculty of Medicine Dursun Odabas Medical Center, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No